CLINICAL TRIAL: NCT04645069
Title: A First-in-Human (FIH), Open-Label, Phase 1/2 Dose Escalation and Expansion Study of ADG126, ADG126 in Combination With Anti PD1 Antibody, and ADG126 in Combination With ADG106 in Patients With Advanced/Metastatic Solid Tumors
Brief Title: ADG126, ADG126 in Combination With Anti PD1 Antibody, and ADG126 in Combination With ADG106 in Advanced/Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adagene Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADG126-1001
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Advanced/Metastatic Solid Tumors
Keywords: Advanced/Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ADG126 mono dose escalation (Experimental): ADG126 monotherapy dose escalation will be traditional 3+3 cohort design.
  Interventions: Biological: ADG126 Mono
- ADG126 mono dose expansion (Experimental): Monotherapy dose expansion is designed to evaluate the preliminary antitumor activity of ADG126 at RP2D or the doses approved by the SRC.
  Interventions: Biological: ADG126 Mono
- ADG126-anti PD1 drug dose escalation (Experimental): Combination therapy will commence at a dose level lower than the cleared dose from the monotherapy dose escalation arms and approved by the SRC.
  Interventions: Biological: ADG126-anti PD1
- ADG126-anti PD1 drug dose expansion (Experimental): Combination therapy expansion will commence at RP2D or the dose approved by the SRC.
  Interventions: Biological: ADG126-anti PD1
- ADG126-ADG106 dose escalation (Experimental): Combination therapy will commence at a dose level lower than the cleared dose from the monotherapy dose escalation arms and approved by the SRC.
  Interventions: Biological: ADG126-ADG106
- ADG126-ADG106 dose expansion (Experimental): Combination therapy expansion will commence at RP2D or the dose approved by the SRC.
  Interventions: Biological: ADG126-ADG106

INTERVENTIONS:
Biological: ADG126 Mono — ADG126 will be administered as an IV infusion over 30-60 minutes ± 15 minutes.
  Arms: ADG126 mono dose escalation; ADG126 mono dose expansion
Biological: ADG126-anti PD1 — ADG126-toripalimab combination regimen will receive of toripalimab 15 to 30 minutes after the end of the ADG126 infusion
  Arms: ADG126-anti PD1 drug dose escalation; ADG126-anti PD1 drug dose expansion
Biological: ADG126-ADG106 — ADG126-ADG106 combination regimen will be receive of ADG106 15 to 30 minutes after the end of the ADG126 infusion
  Arms: ADG126-ADG106 dose escalation; ADG126-ADG106 dose expansion

SUMMARY:
ADG126, ADG126 in Combination with anti-PD1 antibody, and ADG126 in Combination with ADG106 in Patients with Advanced/Metastatic Solid Tumors .

DETAILED DESCRIPTION:
ADG126 is a novel anti-CTLA-4 fully human IgG1 antibody prodrug that is modified with Adagene Safebody technology to control the activation of anti-CTLA4 activity.ADG106 is a fully human ligand-blocking, agonistic anti-CD137 IgG4 mAb which is expected to enhance the activity of activated T cells. The enhanced antitumor efficacy results observed from the preclinical studies of ADG126 in combination with ADG106 or anti-PD-1 provided further support to explore such combinations in clinical settings for better patient responses.

ELIGIBILITY:
Inclusion criteria

1. Adults ≥18 years of age.
2. ECOG performance status 0 or 1.
3. Estimated life expectancy of more than 12 weeks .
4. Patients with advanced or metastatic solid tumors, confirmed by histologically or pathologically documented, who have progressed after all standard therapies, or for whom no further standard therapy exists.
5. At least 1 measurable lesion at baseline according to the definition of RECIST v1.1.
6. Adequate organ function.
7. Meets the additional tumor type requirements as specified in Protocol.

Exclusion Criteria:

1. Treatment with any investigational drug within washout period.
2. Major trauma or major surgery within 4 weeks prior to first dose of study drug(s)
3. History of significant immune-mediated AE.
4. Central nervous system (CNS) disease involvement.
5. Prior organ allograft transplantations or allogeneic peripheral blood stem cell (PBSC)/bone marrow (BM) transplantation
6. Clinically significant cardiac disease.
7. Evidence of active uncontrolled viral, bacterial, or systemic fungal infection.
8. Patients who received:

   1. A COVID-19 vaccine within 7 days of Cycle 1 Day 1.
   2. Live vaccines or live-attenuated vaccines within 28 days prior to Cycle 1 Day 1.
9. Known active infection of HBV/BCV/HIV.
10. Patients requiring systemic treatment with corticosteroids or other immunosuppressive medications (>10 mg/day prednisone or equivalent).
11. Second primary malignancy not in remission for greater than 3 years.
12. History(within the last 5 years) or risk of autoimmune disease.
13. Pregnant or breastfeeding females.
14. Childbearing potential who does not agree to the use of contraception during the treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities escalating dose levels in adults with advanced / metastatic solid tumors | From first dose of ADG126 (Week 1 Day 1) until 21 days
Number of participants with adverse events as assessed by CTCAE v5.0 ADG126-ADG106 combination regimens | From first dose of ADG126 (Week 1 Day 1) to 90 days post last dose

SECONDARY OUTCOMES:
Antidrug antibodies (ADAs) | From first dose (Cycle 1 Day 1, ) until the last dose (up to 2 years)
Area under the time concentration curve (AUC) from time zero to infinity (AUC0-inf) | From first dose (Cycle 1 Day 1, ) until the last dose (up to 2 years)
Maximum (peak) plasma concentration (Cmax) | From first dose (Cycle 1 Day 1, ) until the last dose (up to 2 years)
Time to maximum (peak) plasma concentration (Tmax) | From first dose (Cycle 1 Day 1, ) until the last dose (up to 2 years)
Trough plasma concentration (Ctrough) | From first dose (Cycle 1 Day 1, ) until the last dose (up to 2 years)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - Next oncology, San Antonio, Texas
- Australia (5):
  - Southside Cancer Care Centre, Miranda, New South Wales
  - Macquarie University Hospital, Sydney, New South Wales
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Cabrini Health Limited, Malvern, Victoria
  - One Clinical Research Pty Ltd, Nedlands, Western Australia
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore